CLINICAL TRIAL: NCT06173778
Title: A Randomized Controlled Trial of Once-Weekly Semaglutide for Limiting Post-Smoking Cessation Weight Gain in Adult Smokers With Overweight/Obesity
Brief Title: Semaglutide for Post-Smoking Cessation Weight Management
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Luba Yammine, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-23-0485
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight; Cigarette Smoking
Keywords: smoking; quit smoking; cigarettes; tobacco; overweight; obesity; obesity medications; semaglutide
MeSH Terms: conditions — Obesity; Overweight; Cigarette Smoking; Smoking | interventions — semaglutide; Nicotine Replacement Therapy; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- semaglutide (Experimental)
  Interventions: Drug: semaglutide 2.4mg; Drug: Nicotine Replacement Therapy (NRT, nicotine patch); Behavioral: Brief Smoking Cessation Counseling
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Nicotine Replacement Therapy (NRT, nicotine patch); Behavioral: Brief Smoking Cessation Counseling

INTERVENTIONS:
Drug: semaglutide 2.4mg — Semaglutide 2.4mg will be self-administered once a week under the surface of the skin and will be started at 0.24mg once a week for 4 weeks; in 4-week intervals, the dose will be increased until a dose of 2.4mg is reached
  Arms: semaglutide
Drug: Placebo — Non-active medication, self-administered
  Arms: placebo
Drug: Nicotine Replacement Therapy (NRT, nicotine patch) — Participants who smoke >10 cigarettes/day will use 21 mg patches for the first 6 weeks, 14 mg patches during weeks 7 and 8, and 7 mg patches during weeks 9 and 10. Participants who smoke 5-10 cigarettes per day will use 14 mg patches for the first 6 weeks and 7 mg patches for weeks 7-10.
Behavioral: Brief Smoking Cessation Counseling — Participants will receive weekly, manual-based individual smoking cessation counseling. Counseling will be provided by master's level clinicians.

SUMMARY:
This trial will examine the effect of semaglutide 2.4mg on changes in body weight, body composition, and peripheral and central mechanisms that control appetite, satiety, and food intake in the context of smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent before any study-related activity, willing to comply with al study procedures, and be available for the duration of the study.
* Body mass index (BMI) ≥30 kg/m2 or ≥27 kg/m2 with the presence of at least one of the following weight-related comorbidities (treated or untreated): hypertension (unless meets medical exclusion criterion 7), cardiovascular disease (unless meets medical exclusion criterion 6), dyslipidemia, or obstructive sleep apnea
* Have been smoking ≥5 cigarettes per day for at least 1 year (prior to screening) and provide positive cotinine test.
* Desire to quit smoking (defined as "intend to quit within one month")
* Agree (if the participant is female and of child-bearing potential) to use effective contraceptive methods, unless the participant's male partner(s) is surgically sterile (underwent vasectomy).
* Women of child-bearing potential must provide negative urine pregnancy tests prior to randomization.
* Normal cognitive restraint (assessed as cognitive restraint score of <4 from the Three Factor Eating Habits Questionnaire)
* Have a medical history and a brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the Study Physician and the Principal Investigator

Exclusion Criteria:

Medical Exclusions

* Personal or first-degree relative(s) history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2).
* Acute pancreatitis within the past 6 months prior to screening.
* History or presence of chronic pancreatitis.
* Type 1 or type 2 Diabetes Mellitus (previously diagnosed or indicated by HbA1C ≥48 mmol/mol (6.5%) as measured by central laboratory at screening).
* End stage renal disease (ESRD, previously diagnosed or indicated by estimated glomerular filtration rate (eGFR) value of eGFR < 15 ml/min/1.73 m2 as measured by central laboratory at screening).
* Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischemic attack within the past 60 days prior to screening.
* Systolic blood pressure (SBP) >159 mmHg and/or diastolic blood pressure (DBP) >99 mmHg)
* History of malignant neoplasms within the past 5 years prior to screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed.
* Severe gastrointestinal disease (i.e., severe gastroparesis).
* Known or suspected hypersensitivity to nicotine/nicotine patches; semaglutide, excipients, or related products.
* Women who are currently pregnant, or plan to become pregnant, or lactating, or of childbearing potential and are not using medically accepted forms of contraception.
* Have any illness or condition which in the opinion of the Principal Investigator and/or the Study Physician would preclude safe and/or successful completion of the study.

Psychiatric / Substance Use Exclusions

* Psychoactive substance abuse or dependence (excluding nicotine dependence) within the past 3 months prior to screening (existing diagnosis or as determined by the structured interview).
* Urine drug test positive, before randomization, for any of the following substances:

  1. benzodiazepines
  2. cocaine
  3. opioids
  4. amphetamines
  5. methamphetamine
  6. buprenorphine
  7. barbiturates
  8. 3,4-methylenedioxy-methamphetamine (MDMA)
  9. Tetrahydrocannabinol (THC)
* Psychotic or bipolar disorder, or mood disorder with psychotic features; or eating disorder (existing clinical diagnosis or as determined by the structured interview)
* Moderate to high risk for suicidality (as determined by the structured interview).

Weight-Related Exclusions

* Previously undergone bariatric surgery
* Gained/lost ≥4.5 kg over the past 6 months (prior to screening)
* Currently enrolled in a behavioral weight management plan
* Uncontrolled thyroid disease (the criterion will be assessed at the Study Physician's and the Principal Investigator's discretion)

Smoking-Related Exclusions

-Currently using other combustible (e.g., cigars), other (e.g., chewing tobacco, snuff, snus) or alternative (e.g., electronic cigarettes) tobacco products

Medication-Related Exclusions

* Currently using oral or injectable glucose lowering medications
* Currently using pharmacotherapy for smoking cessation (NRT, varenicline, or bupropion)
* Currently or recently (last 90 days prior to screening) taking medication used for weight management (i.e., orlistat, lorcaserin,vi naltrexone-bupropion, liraglutide, phentermine, topiramate, benzphetamine, diethylpropion, phendimetrazine)
* Currently or recently (within the past 14 days prior to screening) taking medication(s) known to impact appetite and/or weight (i.e., corticosteroids, excluding inhaled)

General Exclusions

* Current, anticipated, or pending enrollment in another research study during this trial that could potentially affect participant safety and/or the study data/design as determined by the Principal Investigator and/or Study Physician.
* Not planning to live in the area for the duration of this trial.
* Surgery scheduled for the duration of the trial, except for minor surgical procedures, in opinion of the Principal Investigator and/or the Study Physician.
* Unable to communicate (read, write, and speak) fluently in English.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Body Weight Percent | Baseline to Week 28

SECONDARY OUTCOMES:
Change in body weight as measured in kilograms (kg) | Baseline to Week 28
Change in body fat mass as measured in kilograms (kg) | Baseline to Week 28
Change in waist circumference as measured in centimeters(cm) | Baseline to Week 28

CONTACTS AND LOCATIONS:
Overall Officials: Luba Yammine, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - The University of Texas at Austin, Austin, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yammine L, Leidy H, Maki KC, Weaver MF, Bodalski EA, Schmitz JM. A randomized controlled trial of once-weekly semaglutide for limiting post-smoking cessation weight gain in smokers with overweight/obesity: Study protocol. Contemp Clin Trials. 2025 Aug;155:107989. doi: 10.1016/j.cct.2025.107989. Epub 2025 Jun 18. PMID 40554081